CLINICAL TRIAL: NCT05236088
Title: The Effects of Neuromuscular Electrical Stimulation in Individuals With Urinary Incontinence After Prostatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, seyda toprak celenay, associate professor, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/02/02
Record Dates: First submitted 2022-02-02; First posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NMES group (Experimental): Neuromuscular electrical stimulation (NMES) will be applied with INNOVO brand (Atlantic Therapeutics, Galway, Ireland) device for 30 minutes 3 days a week during 4 weeks
  Interventions: Device: Neuromuscular electrical stimulation application
- Sham group (Sham Comparator): Sham group will be applied from the same device (INNOVO brand (Atlantic Therapeutics, Galway, Ireland)), for 3 days a week for 30 minutes during 4 weeks, but no current will be given from the device.
  Interventions: Device: Sham neuromuscular electrical stimulation application

INTERVENTIONS:
Device: Neuromuscular electrical stimulation application — It was applied with INNOVO brand (Atlantic Therapeutics, Galway, Ireland) device. It was applied for 30 minutes 3 days a week during 4 weeks
  Arms: NMES group
Device: Sham neuromuscular electrical stimulation application — Sham group will be applied from the same device, again 3 days a week for 30 minutes during 4 weeks, but no current will be given from the device.
  Arms: Sham group

SUMMARY:
The aim of this study is to investigate the effects of neuromuscular electric stimulation on urinary symptoms, quality of life, sexual function, perception of improvement and patient satisfaction in individuals with post-prostatectomy urinary incontinence

DETAILED DESCRIPTION:
One of the two most common complications after prostatectomy surgeries is urinary incontinence (UI) and the other is erectile dysfunction. There are conservative and surgical treatment options in post-prostatectomy urinary incontinence. One of the conservative treatment options is neuromuscular electrical stimulation application. Since electrical stimulation applications, used in the treatment of post-prostatectomy urinary incontinence, are usually given together with other treatment protocols, there are limitations in clearly demonstrating the effects of neuromuscular electrical stimulation on post-prostatectomy urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Being a male individual with stress or stress-dominant mixed urinary incontinence symptoms after undergoing prostatectomy surgery in the urology clinic
* Being over 40 years old
* Volunteering to participate in the study

Exclusion Criteria:

* Severe cardiovascular disease (unstable angina and arrhythmia patients, heart failure patients ect.)
* Those with sensory loss
* Presence of ongoing urinary infection
* Only urgency urinary incontinence
* Having a pacemaker
* Active cancer treatment (radiotherapy, chemotherapy),
* Those who have undergone Transurethral Prostatectomy (TUR-P) surgery
* Those who have a problem that interferes with cooperation and understanding

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male with post-prostatectomy urinary incontinence
Enrollment: 50 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Urinary incontinence severity | change from baseline at 4 weeks
  Urinary incontinence severity will be assess with a 1-hour pad test. This amount; less than 2 grams is considered normal, 2-10 grams is mild, 10-50 grams is moderate, and 50 grams is severe stress urinary incontinence.

SECONDARY OUTCOMES:
Presence of urinary incontinence symptoms | change from baseline at 4 weeks
  Urinary incontinence symptoms will be assessed with International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF). It consists of 6 questions in total and the total score is 3., 4., 5. It is obtained by adding the scores they get from the questions. A low score in the scale indicates that urinary incontinence symptoms are less.
Life quality | change from baseline at 4 weeks
  Life quality will be assessed with King Health Questionnaire. The questionnaire, consisting of thirty-two items, consists of 2 parts. In the first part, there are 2 questions questioning the general health perception and incontinence effect, and 19 questions dividing the quality of life into 7 areas (role limitations, physical limitations, social limitations, personal relationships, emotional problems, sleep/energy disorders, symptom severity measurement). In the second part, there are 11-item complaint severity scales that evaluate the presence and severity of urinary symptoms. While the best score that can be obtained on the complaint severity scale is "0", the worst score is "30", the best score that can be obtained for all King Health Questionnaire subsections is "0" and the worst score is "100".
Sexual function | change from baseline at 4 weeks
  Sexual function will be assessed with International Index of Erectile Function-5. It includes 5 main topics; erectile function, orgasm function, sexual desire, sexual intercourse satisfaction and general satisfaction are questioned with a total of 5 questions. Each question gets a score between 0-5. Total score; severe (5-7), moderate (8-11), mild-moderate (12-16), mild (17-21), no erectile dysfunction (22-25)
Patients' subjective perception of improvement | after treatment (4th week)
  Patients' subjective perception of improvement will be questioned with a 4-point Likert scale (worse (1), same (2), better (3) and completely cured (4)).
Patient satisfaction | after treatment (4th week)
  Patient satisfaction will be questioned with a 5-point Likert scale (not at all satisfied (1), dissatisfied (2), undecided (3), satisfied (4), very satisfied (5))

CONTACTS AND LOCATIONS:
Overall Officials: Seyda Toprak Celenay, Principal Investigator — Ankara Yildirim Beyazıt University